CLINICAL TRIAL: NCT04198207
Title: Clinical Evaluation of the Effectiveness and Safety of Vagus Nerve Stimulation for Tuberous Sclerosis Complex Related Epilepsy
Brief Title: The Effectiveness and Safety of Vagus Nerve Stimulation for TRE
Status: Completed | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); The First Bethune Hospital of Jilin University (Unknown); Xuanwu Hospital, Beijing (Other); Capital Medical University (Other); Peking University First Hospital (Other); China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other); Fourth Medical Center of PLA General Hospital (Other); Capital Institute of Pediatrics, China (Other); The Second Hospital of Hebei Medical University (Other); Xijing Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Children's Hospital of Fudan University (Other); RenJi Hospital (Other); Jining Medical University (Other); Xiamen Humanity Hospital (Other); Xiangya Hospital of Central South University (Other); Wuhan Medical Care Center for Women and Children (Unknown); Guangdong 999 Brain Hospital (Other); Shenzhen Children's Hospital (Other Government); Army Medical University, China (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Shuli Liang, Director of Functional Neurosurgery, Beijing Children's Hospital
Other Study IDs: TRE-VNS
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Tuberous Sclerosis Complex; Epilepsy
Keywords: tuberous sclerosis complex; epilepsy; vagus nerve stimulation
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VNS Group: VNS group: 20 patients with no localilzed epileptogenic tuber in the brain, and with VNS and multiple anti-seizure medicines.
- Control Group: Control group: 50 patients with no localilzed epileptogenic tuber in the brain, and with multiple anti-seizure medicines.

SUMMARY:
Prospective cohort studies to identify clinical epilepsy control, cognitive changes, and safety of VNS in patients with tuberous sclerosis complex-related epilepsy.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of vagus nerve stimulation (VNS) in the treatment of drug-resistant epilepsy in patients with Tuberous Sclerosis Complex (TSC) and compare it with traditional antiepileptic drug therapy. By assessing seizure frequency, severity, and improvements in quality of life, the study seeks to provide evidence-based guidance for clinical treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age Range: Patients aged 1 to 18 years.
* Confirmed Diagnosis: Diagnosed with Tuberous Sclerosis Complex (TSC) according to established diagnostic criteria.
* Drug-Resistant Epilepsy: Ineffectiveness of at least two antiepileptic drugs (monotherapy or combination therapy).
* Informed Consent: Patients and their guardians understand the purpose of the study and voluntarily sign the informed consent form.

Exclusion Criteria：

* Other Severe Diseases: Presence of significant cardiovascular, respiratory, or other systemic diseases.
* Psychiatric Disorders: History or presence of severe psychiatric disorders (e.g., schizophrenia or major depressive disorder).
* Surgical Contraindications: Unsuitability for general anesthesia or factors affecting surgical safety.
* Drug Allergy: Known allergy to drugs used in the study.
* Implant Conflict: Presence of implanted medical devices that may interfere with VNS therapy.
* Pregnancy or Lactation: Pregnant or breastfeeding individuals.
* Poor Compliance: Inability to adhere to follow-up visits or treatment protocols.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from multiple epilepsy centers in China
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
% of patients with Mchugh grading | 4 years
  The grading made by Mchugh for the classification of outcome with respect to epileptic seizures following epilepsy surgery. It contains a total of 5 levels. The higher the level, the worse the result. We will count the percentage of patients at each level.epileptic seizures following epilepsy surgery. It is used for assessing the control of epilepsy.

SECONDARY OUTCOMES:
IQ | 3 years
  Wechsler Intelligence Scale is used for the evaluation of IQ
Quality of Life: QOLIE-31 | 3 years
  QOLIE-31 is suitable for patients 14 years and older. QOLCE-76 is applied to patients aged 2-13 by parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No